CLINICAL TRIAL: NCT03325491
Title: Assessing the Effects of Increased Mitochondrial Function and Chronic Aerobic or Resistance Exercise Training on Skeletal Muscle Performance in Older Men; a Pilot Study
Brief Title: Assessing the Effects of Increased Mitochondrial Function Exercise Training on Muscle Performance
Acronym: Rejuvenate2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges recruiting healthy, sedentary 65-75 year old males
Sponsor: University of Exeter (Other)
Collaborators: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1617/024
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Impaired Mitochondrial Function, Muscle Performance
MeSH Terms: interventions — acipimox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acipimox plus exercise training (Experimental): The active supplement will contain the prescription drug Acipimox (250 mgs) , a nicotinic acid precursor traditionally used to lower blood lipid levels. The supplement will be administered 3 times per day, for 6 weeks.
  Interventions: Dietary Supplement: Acipimox
- Placebo plus exercise training (Placebo Comparator): The placebo supplement will contain only cellulose microcrystalline. This is an inert substance widely used in many pill and tablet formulations. It is an insoluble fibre and is not absorbed into the blood stream therefore is unlikely to cause toxicity when taken orally.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Acipimox — Acipimox plus exercise training: Oral supplement containing Acipimox 250mgs as the active ingredient in blinded label tablet form.
  Arms: Acipimox plus exercise training
Dietary Supplement: Placebo — Alternate unilateral resistance and aerobic exercise training will also be performed 5 times per week for 6 weeks.
  Arms: Placebo plus exercise training

SUMMARY:
As people grow older skeletal muscle gradually becomes smaller and weaker, causing reduced mobility and quality of life. To understand and reverse this negative process investigators need to find new ways of improving the ability of muscle to perform physical activity. There is some evidence that supplements may improve how the mitochondria work, and investigators want to explore this idea in more detail. This is possible by measuring how the muscles work and respond to exercise before and after taking the supplement alongside an aerobic (i.e. cycling) and resistance (i.e. weight lifting) exercise programme. This will give us the basic information investigators would need to see if this is a useful idea.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 65-75 years
* Body mass index between 19-29
* No active cardiovascular or metabolic disease
* No active respiratory disease
* No current musculoskeletal injuries
* A sedentary lifestyle (i.e. does not engage in strenuous, planned physical activity)
* The ability to give informed consent

Exclusion Criteria:

* Currently taking a statin drug or NSAIDs
* Have a current peptic ulcer
* Have any renal impairment
* Have a known hypersensitivity to Acipimox
* Suffer from vertigo
* Smoker

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Change in mitochondrial function | Baseline, 3 weeks, 6 weeks
  Mitochondria will be extracted from muscle samples immediately post-biopsy (biopsies taken baseline, week 3 and week 6) and analysed for content and subsequently for oxidative respiratory function using the Oroboros technique, and maximal rates of Adenosine Triphosphate (ATP) production.

SECONDARY OUTCOMES:
Chronic changes in habitual muscle protein synthetic rates | Baseline, 3 weeks and 6 weeks
  Baseline saliva samples then frequent saliva samples over 6 weeks following oral ingestion of the stable isotope deuterium oxide (D2O, or 'heavy water') will be analysed by gas-chromatography-pyrolysis-isotope ratio mass-spectrometry. analysis. Muscle samples collected at baseline, 3 weeks, 6 weeks will also be analysed by gas-chromatography-pyrolysis-isotope ratio mass-spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Deane, PhD, Principal Investigator — University of Exeter
Locations (1):
- NIHR Exeter Clinical Research Facility, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No